CLINICAL TRIAL: NCT06701721
Title: A Phase 1b Open-Label, Multiple Ascending Dose Study of the Safety, Tolerability, and Biological Activity of Intravitreal THN391 in Diabetic Macular Oedema Secondary to Non-Proliferative Diabetic Retinopathy.
Brief Title: A Study Intravitreal THN391 in Diabetic Macular Oedema Secondary to Non-Proliferative Diabetic Retinopathy.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Therini Bio Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Therini Bio, Inc. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: THN391-OPT-101
Record Dates: First submitted 2024-11-19; First posted 2024-11-22 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Macular Edema; Diabetic Retinopathy
Keywords: Diabetic Macular Oedema; Non-proliferative Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: Multiple Ascending Dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequential Multiple Ascending Doses (Experimental): Participants will be sequentially enrolled to a low, medium, and high doses and receive a total of 3 monthly treatments.
  Interventions: Drug: THN391 MAD

INTERVENTIONS:
Drug: THN391 MAD — Route of administration- IVT injection

SUMMARY:
THN391-OPT-101 is a study assessing safety and preliminary efficacy of THN391 in patients with diabetic macular edema (DME) given as monotherapy.

DETAILED DESCRIPTION:
This is an open label, multiple ascending dose (MAD) study, in which the safety of THN391 will be assessed in escalating doses. This study will enroll a total of approximately 21 participants into 3 sequential dose-escalating cohorts. Participants will receive 3 monthly THN391administrations.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to understand the study procedures and the risks involved and provide written informed consent before the first study-related activity
* 18 to 80 years of age (inclusive at the time of informed consent).
* Diagnosis of Diabetic Macular Edema (DME)
* Vision loss in the study eye

Exclusion Criteria:

* Be pregnant or breastfeeding
* Cataract surgery or any other previous ocular surgery in the study eye within 3 months before Screening
* Any other condition except for DME that could affect interpretation of study assessments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-12-18 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Up to 16 weeks following first dose administration
  Safety and tolerability assessed using ophthalmic examination, imaging, systemic adverse events, and laboratory abnormalities

SECONDARY OUTCOMES:
Change in Visual Acuity | Up to 16 weeks following first dose administration
  Measured using ETDRS method
Change in Retinal Edema | Up to 16 weeks following first dose administration
  Measured with Optical Coherence Tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Naor, Study Director — Therini Bio, Inc.
Locations (2):
- Australia (2):
  - Marsden Eye Specialists, Parramatta, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No